CLINICAL TRIAL: NCT01816997
Title: The Influence of Statins on Glucose Homeostasis and the Biomarkers of Diabetes in Subjects With Impaired Fasting Glucose
Brief Title: The Statins on Glucose Homeostasis in Subjects With Impaired Fasting Glucose
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Principal Investigator, vghtpe user, Taipei Veterans General Hospital, Taipei Veterans General Hospital, Taiwan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: VGHIRB 2011-10-005IA
Record Dates: First submitted 2012-12-28; First posted 2013-03-22 (Estimated); Last update posted 2013-11-18 (Estimated); Status verified 2013-11

CONDITIONS: Diabetes
Keywords: Statins; Glucose homeostasis; Diabetes; Impaired fasting glucose
MeSH Terms: conditions — Diabetes Mellitus | interventions — Pravastatin; Rosuvastatin Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control (Placebo Comparator): IFG subjects with total cholesterol less than 200 mg/dL will be served as controls.
  Interventions: Drug: Control
- Pravastatin (Active Comparator): The impaired fasting glucose (IFG) subjects with total cholesterol 200-280 mg/dL will be randomized into two groups: pravastatin 40 mg or rosuvastatin 10 mg.
  Interventions: Drug: Pravastatin
- Rosuvastatin (Experimental): The impaired fasting glucose (IFG) subjects with total cholesterol 200-280 mg/dL will be randomized into two groups: pravastatin 40 mg or rosuvastatin 10 mg.
  Interventions: Drug: Rosuvastatin

INTERVENTIONS:
Drug: Pravastatin — The impaired fasting glucose (IFG) subjects with total cholesterol 200-280 mg/dL were randomized into two groups: pravastatin 40 mg or rosuvastatin 10 mg.
  IFG subjects with total cholesterol less than 200 mg/dL will be served as controls.
  Other Names: Pravastatin (Mevalotin)
  Arms: Pravastatin
Drug: Rosuvastatin — The impaired fasting glucose (IFG) subjects with total cholesterol 200-280 mg/dL were randomized into two groups: pravastatin 40 mg or rosuvastatin 10 mg.
  IFG subjects with total cholesterol less than 200 mg/dL will be served as controls.
  Other Names: Crestor
  Arms: Rosuvastatin
Drug: Control — placebo
  Other Names: placebo
  Arms: Control

SUMMARY:
Evaluate the effects of rosuvastatin (maybe the highest diabetogenic) and pravastatin (seems to be protective) on the glucose homeostasis and other biomarkers in subjects with impaired fasting glucose.

DETAILED DESCRIPTION:
Statin therapy effectively reduces cardiovascular events. However, trial data1 and meta-analyses suggest that statins also confer increased risk of development of diabetes. In order to elucidate whether statins increase risk of diabetes, investigators conducted this study to evaluate the effects of rosuvastatin (maybe the highest diabetogenic) and pravastatin (seems to be protective) on the glucose homeostasis and other biomarkers in subjects with impaired fasting glucose.

ELIGIBILITY:
Inclusion Criteria:

1. Age 35-70 years old
2. Fasting blood glucose 100-125 mg/dL

Exclusion Criteria:

1. A1C >7.0%
2. 2hr glucose during OGTT >200 mg/dL
3. Total cholesterol >280 mg/dL
4. Previous diabetic history, coronary artery disease
5. Allergy to rosuvastatin or parvastatin
6. Baseline ALT more than 3 times UNL
7. Serum Cr > 2.0 mg/dL
8. Pregnancy, breast feeding or plan to be pregnant woman.

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2012-01; Primary Completion 2017-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Glucose homeostasis | 6 months
  Compare the glucose homeostasis and some biomarkers of diabetes among control, parvastatin and rosuvastatin groups.
  Glucose and insulin response during OGTT. Some markers of insulin resistance and insulin secretion calculated from OGTT.

SECONDARY OUTCOMES:
Some biomarkers of diabetes | 6 months
  Such as GLP-1, GIP, IGF-1, HbA1c, FPG etc.
Progression of glucose homeostasis | 5 to 10 years.
  We will repeat FPG and A1C every 6 months and OGTT every 1-2 years for up to 10 years to investigate the change of these parameters.
Chronic complications of diabetes | Up to 10 years
  Retinopathy: The change of steps on the ETDRS Severity Scales. Nephropathy: UACR and eGFR change. All-cause mortality
Incidence of diabetes | 5 to 10 years.
  We will repeat FPG and A1C every 6 months and OGTT every 1-2 years for up to 10 years to investigate the incidence of diabetes.
Chronic complications of diabetes | Up to 10 years
  Diabetic retinopathy: Development of advanced diabetic retinopathy. Advanced diabetic retinopathy was defined as development of proliferative diabetic retinopathy, retinopathy treated with laser photocoagulation or vitrectomy.
  Nephropathy: Development of macroalbuminuria (UACR >30 mg/mmol creatinine), a severe decline in eGFR (<30 mL/[min•1.73 m2]).
  Cardiovacular events: angina, myocardial infarction, heart failure, acute coronary syndrome and cerebrovascular accident.

CONTACTS AND LOCATIONS:
Overall Officials: Harn-Shen Chen, MD, PhD, Principal Investigator — Taipei Veterans General Hospital, Taiwan
Locations (1):
- Taipei Veterans General Hospital, Taipei, Taipei, Taiwan

REFERENCES:
- [Derived] Cheng WY, Chang LH, Chen HS. The effect of statin treatment on glucose homeostasis in prediabetic individuals: A prospective, randomized, controlled trial. J Chin Med Assoc. 2024 Jul 1;87(7):664-669. doi: 10.1097/JCMA.0000000000001114. Epub 2024 May 29. PMID 38810093